CLINICAL TRIAL: NCT04286334
Title: Three-dimensional Bone Regeneration Using Custom-made Meshes With and Without Collagen Membrane: Randomized Clinical Trial
Brief Title: Three-dimensional Bone Regeneration Using Custom-made Meshes With and Without Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GBR Academy (Network)
Responsible Party: Principal Investigator, Alessandro Cucchi, Principal Investigator, GBR Academy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMF 01/2017
Record Dates: First submitted 2019-02-12; First posted 2020-02-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Surgical Procedure, Unspecified; Soft Tissue Infections; Surgical Wound Dehiscence; Bone Density; Bone Loss in Jaw
MeSH Terms: conditions — Soft Tissue Infections; Surgical Wound Dehiscence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeon is masked until the envelope opening at the end of the surgery, just before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - control Group (Active Comparator): Customized titanium mesh without collagen membrane 15 patients will undergo bone regeneration with custom-made mesh without a collagen membrane. (Meshes - 3D-mesh BTK, Biotec, Vicenza, Italy.) Digitally designed by an operator before the surgery (digital technique).
  Interventions: Device: Bone augmentation with cad-cam laser-sintered mesh
- Group B - Test Group (Experimental): Customized titanium mesh with collagen membrane 15 patients will undergo bone regeneration with a custom-made titanium mesh (BTK, Biotec- Vicenza, Italy). Digitally designed by an operator before the surgery (digital technique), covered by collagen membrane (Cytoplast RTM, Osteogenics, deore materials, Verona, Italy).
  Interventions: Device: Bone augmentation with cad-cam laser-sintered mesh

INTERVENTIONS:
Device: Bone augmentation with cad-cam laser-sintered mesh — Titanium meshes cad cam laser-sintered were applied in sites with alveolar bone deficiency in order to regenerate the bone volume in need of implant-prosthetic restorations.

SUMMARY:
The presence of alveolar ridge deficiencies is considered major limitation to achieve an implant-prosthetic restoration with high aesthetics and stability over time. Guided Bone Regeneration (GBR) can be considered an effective solution for bone augmentation. The most advanced technology of GBR is the customized titanium mesh, which is developed with a fully digital work flow system. The aim of this study is to evaluate complications and bone augmentation rates after GBR, based on customized meshes with or without collagen membranes.

After ethical committee approval, 30 patients with horizontal and/or vertical bone defects were enrolled and treated according to the study protocol. During reconstructive surgery (T0), patients were randomly divided into two study groups: 15 patients were treated by means of a custom-made mesh without collagen membrane (Group A - Control Group), while 15 patients were treated by means of a custom-made titanium mesh with a collagen membrane (Group B - Test Group). All sites were grafted with a mixture 50:50 of autogenous bone and xenograft and primary closures of surgical sites were obtained to ensure a submerged healing of the meshes. After 6 months (T1), re-entry surgery was completed to remove the meshes, evaluate the augmented volume and to place implants in the augmented sites. After 3 months (T2), soft tissue management was accomplished with implant exposure and a connective tissue graft, before prosthetic restoration (T3). Data collection included surgical and healing complications, planned bone volume (PBV) and reconstructed bone volume (RBV), pseudo-periosteum type, bone density, implant success, and crestal bone loss. A statistical analysis of recorded data was performed to investigate any statistically significant differences between the study group and statistical significance was set at a=0.05.

DETAILED DESCRIPTION:
The rationale of the study is based on the fact that manual and intraoperative modeling of an osteosynthesis mesh is an employee operator and even in the case of very experienced operators it is always difficult, inaccurate and slow. The use of this pre-modeled and pre-fabricated custom-made mesh with bevel margins and three-dimensionally morphology adapted to the bone defect, would allow for a congruous bone regeneration reducing the operating times, the risks linked to the mesh trauma, and the discomfort for the patient. The collagen membrane in association with titanium, based on the principles of guided bone regeneration (GBR), would make it possible to increase bone gain and reduce the percentage of early and late exposure of the mesh.

This study aims to evaluate, in cases of maxillary and mandibular atrophies characterized by a vertical and / or horizontal resorption of the alveolar bone, the percentage of complications (intra- and post-operative) after bone regeneration using custom-made mesh with or without collagen membrane.

The primary objective of this study is to evaluate the non-inferiority of technique B (custom-made mesh - without membrane) compared to technique A (custom-made mesh - with membrane) in the incidence of complications.

Secondary objectives include evaluation of the missing bone volume (lacking bone volume or LBV), reconstructed bone volume (reconstructed bone volume or RBV) with respect to planned bone volume (planned bone volume or PBV), histological and histomorphometric analysis at the time removal of the mesh and peri-implant bone resorption, due to the functional loading of the implants, at 12 months of follow-up.

Other objectives include the qualitative evaluation of bone regeneration by histological and histomorphometric analysis upon removal of the mesh; and the evaluation of peri-implant bone resorption, due to the functional loading of the implants, at 12 months of follow-up.

This is a clinical trial which is promoted by Prof. Claudio Marchetti and the University Hospital of Bologna - Policlinico Sant'Orsola Malpighi. The study is designed as a pilot, randomized, monocentric, independent, parallel-group clinical trial, in which the variables will be analyzed prospectively.

The study will have a selection and enrollment period of approximately 12 months; a treatment period of about 12 months. As a result, the overall duration of the study will be around 24 months.

In the two-year period 2017/2019 the study will include the treatment of 30 patients, in good general health, suffering from partial edentulism of the maxilla and / or jaw with vertical and / or horizontal resorption of the alveolar bone, which require prosthetic rehabilitation supported by implants to improve function and aesthetics of edentulous areas.

Patients will be divided into 2 study groups and assigned to each study group based on the previously computer-generated randomization sequence: 15 patients (group A, control) will be treated by bone regeneration with custom-made mesh without a collagen membrane. 15 patients (group B, test) will be treated by bone regeneration with custom-made mesh with collagen membrane.

In the following table, the 3 treatment phases: The first phase (T0) involved bone regeneration with a custom-made mesh (group A) and with collagen membrane (group B); the second one (T1), subsequently, after 6 months: will forsee the removal of the regeneration device and the insertion of the implants; the thirt (T2), 3 months after the aforementioned, will forsee the final functional loading of the implants, with a consequent follow-up of the regenerated bone.

All the materials and tools that will be used in the study are CE certified (with the exception of the custom-made mesh which, as a custom-made device, does not require CE certification) and have already been used in the normal care path for patients who have undergone bone regeneration. Moreover, the control visits and the radiological investigations of the data foreseen by the aforementioned protocol will be collected; They will be summarized in the case report form (CRF), and are those that characterize the normal care path of patients undergoing necessary bone regeneration for prosthetic implant rehabilitation when the bone quantity is insufficient.

The primary objective of this study is to evaluate the non-inferiority of technique B (digital technique) compared to technique A (traditional technique) in the incidence of complications.

The Secondary objectives include: assessment of patient and operator benefits, reconstructed bone volume (RBV) compared to planned bone volume (PBV), histological and histomorphometric analysis of bone quality obtained and peri-implant bone resorption after 12 months of follow-up.

The sample size necessary to support the null hypothesis is 17 subjects for each group. In order to compensate for any protocol deviations or possible drop-outs, the number of patients was increased to 15 per group.

The results obtained in the two study groups will be subjected to descriptive statistical analysis and the differences between groups will be tested by means of appropriate statistical tests for purely exploratory and non-demonstrative purposes.

The patient will be considered as the statistical unit of the analysis, and the statistical significance will be set at α = 0.05.

The collected data will be grouped and summarized with respect to the demographic, anamnestic, and clinical variables of each patient.

Exploratory analyses will be performed using descriptive statistics. The data will be presented both for the intent-to-treat population and for the per-protocol population.

The sample size necessary to support the null hypothesis is 17 subjects for each group. In order to compensate for any protocol deviations or possible drop-outs, the number of patients was increased to 15 per group. The sample size was calculated using dedicated statistical software (STATA, StataCorp LLC) through Pearson's chi-squared test, guaranteeing a level of significance of 95% and a power of 80%.

ELIGIBILITY:
Adult patients, over the age of 18, in good general health.

* Patients with partial edentulism of the maxilla or mandible, with a 2mm minimum to a 12mm maximum vertical bone defect, which requires a three-dimensional bone regeneration intervention in order to have a fixed implant supported rehabilitation.
* Obtaining informed consent for experimental treatment and processing the personal data.

Exclusion Criteria:

* Poor oral hygiene,
* Untreated periodontal disease
* Smoking habit> 10 cigarettes / day;
* Abuse of alcohol or drugs
* Pregnancy
* Patients with odontostomatological infections and / or systemic infections in progress;
* Patient with uncontrolled diabetes mellitus or other metabolic diseases;
* Patients with severe changes in liver and kidney function.
* Patients with confirmed uncontrolled autoimmune disorders.
* Patients subjected radiation therapy in the head or neck region in the last 5 years.
* Patients undergoing immunosuppressive and / or immunocompromised therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The rate of healing complications after reconstructive surgery | 6 months
  Healing complications are evaluated based on the chronological order in which they occur:
  * immediate exposure occurs within the 1st month
  * early exposure occurs between the 1st and the 3rd month
  * late exposure occurs after the 3rd month
  Evaluation of low-grade and high-grade infection of medical devices used for bone regeneration.
  The former complications are classified as:
  * Class A, including flap damage (soft tissue perforation or laceration)
  * Class B, including neurological damage (paresthesia or disesthesia)
  * Class C,including vascular damage (hemorrhage).
  The latter complications are divided into four classes, according to the presence and extent of exposure, as well as the presence of a purulent exudate:
  * Class I, membrane exposure <3 mm, no purulent exudate
  * Class II membrane exposure >=3mm, no purulent exudate
  * Class III: membrane exposure, with purulent exudate

SECONDARY OUTCOMES:
Level of anxiety of the patient measured with a Visual Analogue Scale (VAS) | Immediately before/after surgery
  Level of anxiety measured with a Visual Analogue Scale (VAS), where 0 represents the absence of anxiety and 10 represents the maximum level of anxiety.
Pain level of the patient measured on a Visual Analogue Scale (VAS) | Post operative from immediately after surgery to the 14th day after the surgery
  Pain level measured on a Visual Analogue Scale (VAS), where 0 represents the absence of pain and 10 represents the maximum level of pain.
Total Number of painkillers taken post-operative | Post operative from immediately after surgery to the 14th day after the surgery
  Total amount of pain killers taken from post operative to the 14th day (a two week period) which will be recorded in the patient's diary.
Dosage of painkillers | Post operative from immediately after surgery to the 14th day after the surgery
  Dosage of painkillers measured as the number of painkillers per day, which will be reported in a diary by the patients.
Limitation in daily functions measured on a Visual Analogue Scale (VAS) | Post operative from immediately after surgery to the 14th day after the surgery
  Limitation in daily functions measured on a Visual Analogue Scale (VAS), where 0 represents the absence of limitations and 10 represents the total limitation.
Number of patients' post-operative signs and symptoms | From the 1st day to the 14th day after the surgery.
  Self-assessment of patient's post-operative signs and symptoms (absence or presence swelling, nausea, hematoma, bruising, bleeding), which will be reported in a diary by the patients.
Discomfort level of the patient using a Post-operative Symptom Severity (PoSSe) | Post operative, measured on 14th day after the surgery]
  Discomfort level measured using a Post-operative Symptom Severity (PoSSe) questionnaire.
  Questions are a forced choice, requiring the respondent to tick one box.
  The questions evaluate the discomfort level in different areas:
  * eating: ability to eat, ability to swallow, enjoyment of food, altered taste sensation;
  * speech: voice affected, inability to open mouth, speech affected
  * sensation: tingling of lips or tongue, numbness of lips or tongue
  * appearance: bruising of face and/or neck, swelling of face and/or neck, life affected by appearance
  * pain: days of pain, pain controlled by painkillers, life affected by pain
  * sickness: days of nausea and vomiting, number of attacks of nausea and vomiting on worst day
  * interference with daily activities: interference with work/housework/daily activities, interference with leisure activities
Level of satisfaction of the patient using a Health-Related Quality of Life (HrQoL) | 6 months and 12 months after the dental prosthesis dental prosthesis has been placed.
  Level of satisfaction measured using a Health-Related Quality of Life (HrQoL) questionnaire. Each of the questions are answered with the options of "I am quite satisfied, I'm satisfied, I have no idea, I am dissatisfied, and I am quite dissatisfied".
  The questions evaluate:
  * satisfaction with the overall treatment chewing ability
  * cleaning of the prothesis
  * esthetics of the prothesis
  * speaking ability
Willingness of the patient to undergo the intervention recorded on a Visual Analogue Scale (VAS) | Post operative measured on the 7th day and on the 14th day
  Willingness to undergo the intervention recorded on a Visual Analogue Scale (VAS) where 0 corresponds to "I will never undergo this type of surgery again" and 10 corresponds to "no problem repeating surgery if necessary".
Time required for the CBCT analysis and design of the medical device | Pre-operative, 2 weeks before the day of the surgery
  Time required for the CBCT analysis and design of the medical device measured in a total number of minutes.
Total operative time required for the surgery, measured from immediately before to immediately after the surgery. | During procedure
  Total operative time measured from the time of incision to the end of the suture.
Total chair time measured from immediately before the surgery to immediately after the surgery. | During procedure
  Total chair time measured from the time the patient enters the surgery to the time the patient leaves the room.
Level of operator satisfaction Measured on a 5 point scale | Immediately after the surgery
  Level of operator satisfaction rated on a 5-point scale, ranging from "absolutely not satisfied" to "absolutely satisfied".
Level of operator confidence with the technique | During procedure
  Confidence level with the technique used on a 5-point rating scale, ranging from "absolutely not confident" to " absolutely confident".
Costs related to the technique | Immediately after the surgery
  Costs related to the GBR technique measured as the total costs of the materials used: number of pins, number of screws, number of membranes, number of biomaterials, number of sutures.
Operator anxiety level recorded on a Visual Analogue Scale (VAS) | From 3 days before the surgery to immediately before the surgery, during the intervention and at the 14th day after the surgery.
  Operator anxiety level recorded on a Visual Analogue Scale (VAS), where 0 represents the absence of anxiety and 10 represents the maximum level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Corinaldesi, MD, DDS, MS, Study Director — school of dentistry - University of Bologna
Locations (1):
- School of Dentistry - University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Original articles in international journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From May 2020
Access Criteria: Access credentials to journal resources